CLINICAL TRIAL: NCT00690755
Title: Defective Atypical PKC Activation in Diabetes and Metabolic Syndrome
Brief Title: Defective Atypical Protein Kinase C (PKC) Activation in Diabetes and Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ENDA-037-04F
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetic
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Muscle biopsies taken before and after insulin stimulation in euglycemic clamp studies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Group 1: type 2 diabetic individuals
- Group 2: type 1 diabetic individuals or those with diabetes secondary to pancreatic disease
- Group 3: non-diabetic individuals who are not considered to be overweight
- Group 4: non-diabetic individuals who are considered to be overweight
- Group 5: non-diabetic and type 2 diabetic individuals who will be subjected to an exercise study
- Group 6: individuals who have or are suspected of having glucose intolerance, including patients who have a history of gestational diabetes and patients who have polycystic ovary syndrome
- Group 7: healthy non-diabetic subjects who will receive one dose of metformin orally 1-2 hours before performing procedures

SUMMARY:
The investigators are examining the activation of insulin signaling factors in skeletal muscles of human diabetics. The investigators are characterizing the defects in signaling, and are examining the effects of anti-diabetic agents and exercise on signaling to glucose transport biochemical machinery and whole body glucose disposal.

DETAILED DESCRIPTION:
We have provided clear evidence that insulin activation of all three signaling components, Viz., IRS-1-dependent PI 3-Kinase, atypical protein kinase C (aPKC) and PKB/Akt is defective in diabetic muscle. These defects are best seen when insulin activation is conducted at both half-maximal and maximal stimulation. Moreover, whereas previous studies had shown that treatment with metformin (Met) alone improves aPKC activation, or that treatment with thiazolidinedione (TZD) alone produces increases in activation of IRS-1/PI3K and aPKC when evaluated at maximal insulin stimulation, we have recently found that combined treatment with Met plus TZD for 6 weeks provokes marked increases in insulin effects on all three signaling factors at both half-maximal and maximal insulin stimulation. This work is being prepared for submission for publication.

We have also evaluated the improvement in insulin signaling in diabetic muscle 4 hours after acute endurance (one-legged) exercise and found that the responsiveness of aPKC to the lipid PI3K-derived activator, PIP3, was improved. Also increased was the activation by insulin of IRS-2-dependent PI3K, ERK1/2, and downstream protein synthesis machinery, viz., p70S6 kinase and eukaryotic elongation factor eEF2. These effects of exercise would be expected to enhance glucose transport and utilization by muscle, and promote protein synthesis, i.e., an anabolic response.

ELIGIBILITY:
Inclusion Criteria:

* Stable uncomplicated type 2 diabetes
* Able to be off oral treatments for 2 months

Exclusion Criteria:

* Diabetic complications related to heart, eye, nerve problems
* Renal impairment
* Cardiovascular disease
* Hepatic disease
* Prior history of other disorders or complications caused by diseases
* Insulin therapy needed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes controlled by diet or oral agents and comparable non-diabetic control subjects
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2000-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert V Farese, MD, Principal Investigator — VA Medical Center
Locations (1):
- VA Medical Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as data is presented in the published paper as a mean plus or minus SEM.

REFERENCES:
- [Result] Temofonte N, Sajan MP, Nimal S, Pastoor T, Fumero C, Casaubon L, Powe JL, Standaert ML, Farese RV. Combined thiazolidinedione-metformin treatment synergistically improves insulin signalling to insulin receptor substrate-1-dependent phosphatidylinositol 3-kinase, atypical protein kinase C and protein kinase B/Akt in human diabetic muscle. Diabetologia. 2009 Jan;52(1):60-4. doi: 10.1007/s00125-008-1180-z. Epub 2008 Oct 30. PMID 18972094
- [Result] Beeson M, Sajan MP, Daspet JG, Luna V, Dizon M, Grebenev D, Powe JL, Lucidi S, Miura A, Kanoh Y, Bandyopadhyay G, Standaert ML, Yeko TR, Farese RV. Defective Activation of Protein Kinase C-z in Muscle by Insulin and Phosphatidylinositol-3,4,5,-(PO(4))(3) in Obesity and Polycystic Ovary Syndrome. Metab Syndr Relat Disord. 2004 Spring;2(1):49-56. doi: 10.1089/met.2004.2.49. PMID 18370676
- [Result] Casaubon L, Sajan MP, Rivas J, Powe JL, Standaert ML, Farese RV. Contrasting insulin dose-dependent defects in activation of atypical protein kinase C and protein kinase B/Akt in muscles of obese diabetic humans. Diabetologia. 2006 Dec;49(12):3000-8. doi: 10.1007/s00125-006-0471-5. Epub 2006 Oct 7. PMID 17028898
- [Result] Luna V, Casauban L, Sajan MP, Gomez-Daspet J, Powe JL, Miura A, Rivas J, Standaert ML, Farese RV. Metformin improves atypical protein kinase C activation by insulin and phosphatidylinositol-3,4,5-(PO4)3 in muscle of diabetic subjects. Diabetologia. 2006 Feb;49(2):375-82. doi: 10.1007/s00125-005-0112-4. Epub 2006 Jan 5. PMID 16395615
- [Result] Beeson M, Sajan MP, Dizon M, Grebenev D, Gomez-Daspet J, Miura A, Kanoh Y, Powe J, Bandyopadhyay G, Standaert ML, Farese RV. Activation of protein kinase C-zeta by insulin and phosphatidylinositol-3,4,5-(PO4)3 is defective in muscle in type 2 diabetes and impaired glucose tolerance: amelioration by rosiglitazone and exercise. Diabetes. 2003 Aug;52(8):1926-34. doi: 10.2337/diabetes.52.8.1926. PMID 12882907

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Type 2 diabetic
- Group 2: Type 1 diabetic
- Group 3: Control (non-diabetic)
- Group 4: Non-diabetic overweight
- Group 5: Non-diabetic and Type 2 diabetic
- Group 6: Impaired glucose tolerance (IGT)
- Group 7: Non-diabetic treated with Metformin
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Started | 30 | 0 | 97 | 20 | 0 | 10 | 0
Completed | 28 (Patient recruitment ended on 12/31/2010) | 0 | 51 | 15 | 0 | 6 | 0
Not Completed | 2 | 0 | 46 | 5 | 0 | 4 | 0
Not completed — Physician Decision | 2 | 0 | 46 | 5 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 5: Non-Diabetic and Type 2 Diabetic subjected to exercise study
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Total
Number analyzed (Participants) | 28 | 0 | 51 | 15 | 0 | 6 | 0 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (1) |  | 47 (3) | 51 (3) |  | 43 (3) |  | 47 (4)
Gender [Number; unit: participants]
  Female | 6 |  | 18 | 10 |  | 3 |  | 37
  Male | 22 |  | 33 | 5 |  | 3 |  | 63
Region of Enrollment [Number; unit: participants]
  United States | 28 |  | 51 | 15 |  | 6 |  | 100

OUTCOME MEASURES:

1. Primary Outcome: Alterations in PKC-zeta mRNA in Vastus Lateralis Skeletal Muscles
Description: All muscle samples obtained by 9/30/07, final date for examination of samples 9/30/08 Muscle dependent ability to diminish blood glucose levels during insulin treatment.
Time Frame: PKC-zeta mRNA levels and aPKC activity in muscle evaluated 40 minutes post-insulin treatment
Population: PKC-zeta mRNA and aPKC activity in vastus lateralis skeletal muscle was measured by analysis of gene expression levels of PKC and measuring them in relative amounts in comparison to control subjects.
Measure: Mean (Standard Error); unit: arbitrary units/ng rRNA
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 28 | 0 | 51 | 15 | 0 | 6 | 0
arbitrary units/ng rRNA | 1.76 (0.088) |  | 3.58 (0.179) | 2.14 (0.107) |  | 2.22 (0.110) |
Statistical Analysis 1: Comparison: Group 1 vs Group 3 vs Group 6; Test type: Superiority or Other; p = .001, ANOVA

ADVERSE EVENTS:
Groups:
- Group 1: Diabetics
- Group 2: Type 1 diabetes
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/0 | 0/97 | 0/20 | 0/0 | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 2/30 | 0/0 | 0/51 | 0/15 | 0/0 | 0/6 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=30) | Group 2 (N=0) | Group 3 (N=51) | Group 4 (N=15) | Group 5 (N=0) | Group 6 (N=6) | Group 7 (N=0)
Syncopal event (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
As the study progressed, it was determined that there was not scientific merit to the Groups 2, 5 or 7. These groups were, therefore, not pursued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No